CLINICAL TRIAL: NCT02420639
Title: Prospective, Interventional Study Evaluating the Feasibility and Safety of the Esophageal Cooling Device in 15 Patients Suffering From Traumatic Brain Injury and Treated With Targeted Temperature Management
Brief Title: Prospective, Interventional Study Evaluating the Feasibility and Safety of the Esophageal Cooling Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Cooling Therapy, Inc., d/b/a Attune Medical (Industry)
Collaborators: Dnipropetrovsk State Medical Academy (Other)
Responsible Party: Sponsor
Organization: Advanced Cooling Therapy LLC, d/b/a Attune Medical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ACT TBI-01
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): The placement of the Esophageal Cooling Device will follow standard recommendations as per Instructions for Use. The Esophageal Cooling Device will be connected to the appropriate console (Meditherm III, Blanketrol II, or Blanketrol III).
  Interventions: Device: Esophageal Cooling Device (ECD), manufactured by Advanced Cooling Therapy, Inc.

INTERVENTIONS:
Device: Esophageal Cooling Device (ECD), manufactured by Advanced Cooling Therapy, Inc. — Use of the Esophageal Cooling Device for control of patient temperature.

SUMMARY:
The aim of this prospective, interventional study is to assess the feasibility and safety of the Esophageal Cooling Device in patients from suffering from traumatic brain injury who the treating physician is treating with targeted temperature management. Comparison of outcomes will be made to historical controls. The primary outcome is the feasibility of inducing, maintaining, and rewarming patients from targeted temperature management using the Esophageal Cooling Device (cooling rate, rewarming rate, and the percent of time within goal temperature during the goal-temperature maintenance period). Evaluation of adverse events (including cardiac arrhythmias, severe bradycardia, myocardial infarction/re-infarction, dysphagia, odynophagia, aspiration pneumonia, non-aspiration pneumonia, reflux, esophageal injury, and esophagitis) will be closely monitored during the whole period of targeted temperature management (secondary endpoint).

DETAILED DESCRIPTION:
Controlling patient's body temperature, and in particular, reducing body temperature in a treatment referred to as targeted temperature management, has been shown to improve outcomes for many conditions, including neonatal hypoxic ischemic encephalopathy, cardiac arrest, and traumatic brain injury. However, available modalities for inducing targeted temperature management have a number of technical, logistical, and financial barriers. The Esophageal Cooling Device is a multi-chambered silicone tube placed in the esophagus that provides a highly efficient heat transfer to or from a patient.

Traumatic brain injury (TBI) is a major cause of death and severe disability throughout the world. Current methods of traumatic brain injury treatment include reduction of brain swelling and edema, both by surgical means, as well as by reduction of temperature and avoidance of fever. Methods used to reduce temperature and control fever include surface devices, such as ice packs and water circulating blankets, and intravascular catheters, which are placed into a blood vessel.

The esophagus is in close proximity to blood flow from the heart and great vessels, and the Esophageal Cooling Device (ECD) is designed to take advantage of this heat exchange environment. The ECD's ability to decompress the stomach and avoid distention of the esophagus away from the device ensures good contact with the esophageal mucosa, and thus maximizes heat transfer from the patient. The ECD replaces the standard gastric tube which is placed in the target patient population as a routine standard of care, is made of standard medical-grade silicone, and is generally similar in size and shape to the gastric tubes currently used. Initial mathematical, animal, and human data have shown strong support for the efficacy and safety of the ECD.

The aim of this prospective, interventional study is to assess the feasibility and safety of the Esophageal Cooling Device in patients from suffering from traumatic brain injury who the treating physician is treating with targeted temperature management. Comparison of outcomes will be made to historical controls. The primary outcome is the feasibility of inducing, maintaining, and rewarming patients from targeted temperature management using the Esophageal Cooling Device (cooling rate, rewarming rate, and the percent of time within goal temperature during the goal-temperature maintenance period). Evaluation of adverse events (including cardiac arrhythmias, severe bradycardia, myocardial infarction/re-infarction, dysphagia, odynophagia, aspiration pneumonia, non-aspiration pneumonia, reflux, esophageal injury, and esophagitis) will be closely monitored during the whole period of targeted temperature management (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Patient population will consist of 15 patients suffering from traumatic brain injury, in whom the treating clinician has determined that targeted temperature management will be initiated.

Exclusion Criteria:

* Patients with known esophageal deformity or evidence of esophageal trauma (for example, known esophageal varices, cirrhosis, history of esophagectomy, previous swallowing disorders, achalasia, etc.).
* Patients with known ingestion of acidic or caustic poisons within the prior 24 hours.
* Patients with less than 40 kg of body mass.
* Patients known to be pregnant.
* Terminal disease or "do not resuscitate order" that could lead to early-onset therapeutic withdrawal.
* Unstable hemodynamic conditions that could lead to multi-organ failure and early-onset death.
* Pre-existing severe conductive disorder requiring pacing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleksandr Tsarev, MD, Principal Investigator — Dnipropetrivsk State Medical Academy based on Dnipropetrivsk Regional Clinical Hospital n.a. Mechnikov, Department of Anesthesiology and Intencive Care Medicine, 14 Octoberskay sq., Dnipropetrivsk 49600, Ukraine
Locations (1):
- Dnipropetrivsk State Medical Academy based on Dnipropetrivsk Regional Clinical Hospital, Dnipro, Ukraine

REFERENCES:
- [Background] Arrich J, Holzer M, Havel C, Mullner M, Herkner H. Hypothermia for neuroprotection in adults after cardiopulmonary resuscitation. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD004128. doi: 10.1002/14651858.CD004128.pub3. PMID 22972067
- [Background] Crossley S, Reid J, McLatchie R, Hayton J, Clark C, MacDougall M, Andrews PJ. A systematic review of therapeutic hypothermia for adult patients following traumatic brain injury. Crit Care. 2014 Apr 17;18(2):R75. doi: 10.1186/cc13835. PMID 24742169
- [Background] Andrews PJ, Sinclair LH, Harris B, Baldwin MJ, Battison CG, Rhodes JK, Murray G, De Backer D; Eurotherm3235Trial collaborators. Study of therapeutic hypothermia (32 to 35 degrees C) for intracranial pressure reduction after traumatic brain injury (the Eurotherm3235Trial): outcome of the pilot phase of the trial. Trials. 2013 Sep 3;14:277. doi: 10.1186/1745-6215-14-277. PMID 24004918
- [Background] Polderman KH. Induced hypothermia and fever control for prevention and treatment of neurological injuries. Lancet. 2008 Jun 7;371(9628):1955-69. doi: 10.1016/S0140-6736(08)60837-5. PMID 18539227
- [Background] Badjatia N. Hyperthermia and fever control in brain injury. Crit Care Med. 2009 Jul;37(7 Suppl):S250-7. doi: 10.1097/CCM.0b013e3181aa5e8d. PMID 19535955
- [Background] Kulstad E, Metzger AK, Courtney DM, Rees J, Shanley P, Matsuura T, McKnite S, Lurie K. Induction, maintenance, and reversal of therapeutic hypothermia with an esophageal heat transfer device. Resuscitation. 2013 Nov;84(11):1619-24. doi: 10.1016/j.resuscitation.2013.06.019. Epub 2013 Jul 1. PMID 23827887
- [Background] Markota A, Kit B, Fluher J, Sinkovic A. Use of an oesophageal heat transfer device in therapeutic hypothermia. Resuscitation. 2015 Apr;89:e1-2. doi: 10.1016/j.resuscitation.2015.01.032. Epub 2015 Feb 7. No abstract available. PMID 25660954

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 12 (Study obtained 12 patients)
Completed | 12 (Total of 12 patients enrolled)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Ukraine | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Time to Initiation of Temperature Management
Description: Time to initiation of targeted temperature management, as measured from the time a decision is made to begin targeted temperature management, to the time the esophageal cooling device is in place.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Intervention
Number analyzed (Participants) | 12
hours | 5.83 (5)

2. Secondary Outcome: Composite of Performance Outcomes
Description: Secondary performance outcomes include the feasibility of inducing, maintaining, and rewarming patients from targeted temperature management using the Esophageal Cooling Device. Specifically, cooling rate, rewarming rate, and the percent of time during the goal- temperature maintenance period within 1°C of goal temperature (typically 33°C, but with some centers using anywhere from 32°C to 36°C) will be measured.
Time Frame: 36 hours
Reporting Status: Not Posted

3. Secondary Outcome: Composite of Safety Outcomes
Description: Secondary safety outcomes include evaluation of adverse events including the following: cardiac arrhythmias, severe bradycardia, myocardial infarction/re-infarction, dysphagia, odynophagia, aspiration pneumonia, non-aspiration pneumonia, reflux, esophageal injury, and esophagitis.
Time Frame: Assessed over 36 hours of treatment and up to 30 days of follow-up.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Intervention: The placement of the Esophageal Cooling Device will follow standard recommendations as per Instructions for Use. The Esophageal Cooling Device will be connected to the appropriate console (Meditherm III, Blanketrol II, or Blanketrol III).
  Esophageal Cooling Device (ECD), manufactured by Advanced Cooling Therapy, Inc.: Use of the Esophageal Cooling Device for control of patient temperature. Adverse events specifically monitored included the following: cardiac arrhythmias, severe bradycardia, myocardial infarction/reinfarction, dysphagia, odynophagia, aspiration pneumonia, nonaspiration pneumonia, reflux, esophageal injury, and esophagitis.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=12)
a small volume left hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT02420639/Prot_SAP_000.pdf